CLINICAL TRIAL: NCT01999166
Title: Phenotype/Genotype Correlation in a Family With Early Onset Osteoarthritis: Contribution of Genetic in the Diagnosis and Early Management of Patients.
Brief Title: Phenotype/Genotype Correlation in a Family With Early Onset Osteoarthritis
Acronym: Exorhum
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-A00211-4
Record Dates: First submitted 2013-11-14; First posted 2013-12-03 (Estimated); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — X-Rays

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Osteoarthritis
  Interventions: Radiation: radiography (X-ray); Genetic: DNA sampling

INTERVENTIONS:
Radiation: radiography (X-ray)
Genetic: DNA sampling

SUMMARY:
This study will investigate the genes responsible for osteoarthritis. Individuals with osteoarthritis known or suspected to be caused by a gene mutation (change) may be eligible for this study. Family members may also participate.

Patients will talk with investigators who will explain the study and its possible implications for the patient and family and answer questions. The patient's medical records will be reviewed, a personal and family history will be taken, and a physical examination will be done. Two procedures may be done including blood sampling (which will be used for DNA (genetic) studies) and X-rays (to define osteoarthritis grade).

If no known mutations responsible for osteoarthritis will be detected, participating family members will be interviewed by telephone about their personal and family health history and will have a blood sample drawn for DNA testing, and X-rays.

DETAILED DESCRIPTION:
We will investigate the clinical manifestations and molecular genetic defects of human osteoarthritis. Families with osteoarthritis of known or suspected genetic basis will be enrolled. Individuals will undergo clinical assessment and genetic analyses for the purpose of: 1) definition and characterization of phenotype, 2) determination of the natural history of the disorder, and 3) genotype/phenotype correlation. Genetic linkage studies may be performed for disorders in which the genetic bases is not yet known.

ELIGIBILITY:
Inclusion Criteria:

* Individuals (and family members) with early onset osteoarthritis according to the following definition:

  * symptomatic OA before 50 years old
  * no obvious causes of OA (IMC > 30, dysplasia,joint traumas)
  * at least three OA locations

Exclusion Criteria:

* Individuals younger than 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Family With Early Onset Osteoarthritis
Sampling Method: Non-Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2014-10-07 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Identification of new gene mutations associated with early onset of osteoarthritis using NGS (Next Generation Sequencing) | time of inclusion = Day 0
  Clinical, genetic and imaging factors of osteoarthritis

CONTACTS AND LOCATIONS:
Overall Officials: Christian MARCELLI, Principal Investigator — University Hospital, Caen
Locations (1):
- CHU, Caen, France, France